CLINICAL TRIAL: NCT06007248
Title: Disease Characteristics of Inflammation-associated Rapidly-progressive Coronary Artery Disease (IR-CAD): a Case-control Study
Brief Title: Disease Characteristics of IR-CAD: a Case-control Study
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, LiuZhenyu, Professor, Peking Union Medical College Hospital
Other Study IDs: K3819
Record Dates: First submitted 2023-07-07; First posted 2023-08-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Coronary Artery Restenosis; Coronary Artery Disease Progression; Inflammation; Inflammatory Disease; Inflammation Vascular
Keywords: Coronary Artery Disease; Coronary Revascularization; Progression, Disease; Inflammation; Characteristics Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis; Inflammation; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be retained for exploratory tests, including RNA sequencing, proteomics, and metabolomics, et al.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: IR-CAD patients (from the IR-CAD cohort study)
  Interventions: Diagnostic Test: Protocol-defined Examinations
- Control Group: AS-CAD patients
  Interventions: Diagnostic Test: Protocol-defined Examinations

INTERVENTIONS:
Diagnostic Test: Protocol-defined Examinations — Lab tests (blood and urine and stool routine tests, hepatic and renal and thyroid function tests, tests for metabolic markers, tests for cardiac biomarkers, thrombosis-related tests, rheumatology tests, tests for inflammation markers), electrocardiography, echocardiography, Birmingham Vasculitis Activity Score (BVAS-3), 6-minute walk test, 1-minute squat test, vascular ultrasound, fibroblast activation protein inhibitor (FAPI) positron emission tomography/computed tomography (PET/CT), coronary angiography, optical coherence tomography (OCT), tests for exploratory biomarkers.

SUMMARY:
The present case-control study is designed to investigate the disease characteristics of IR-CAD by comparing the demographics, clinical features, lab results, imaging findings, and prior treatment between 20 patients with IR-CAD and 10 patients with AS-CAD.

DETAILED DESCRIPTION:
A special type of coronary artery disease (CAD) has been identified in the investigators' clinical practice, which has completely different clinical features from those of typical atherosclerotic coronary artery disease (AS-CAD). The patients often have sterile inflammatory diseases and/or clinical evidence of inflammation, whose CAD progresses rapidly, recurs frequently, and responds poorly to intensified secondary prevention of AS-CAD, especially after percutaneous coronary intervention (PCI). The investigators name this special type of CAD with inflammation-associated rapidly-progressive coronary artery disease (IR-CAD). Currently, the overall disease characteristics of IR-CAD remain unknown.

The present case-control study is designed to investigate the disease characteristics of IR-CAD by comparing the demographics, clinical features, lab results, imaging findings, and prior treatment between 20 patients with IR-CAD and 10 patients with AS-CAD.

The first 20 patients who were enrolled in the IR-CAD cohort study, which included patients who met the inclusion/exclusion criteria for IR-CAD and received comprehensive treatment, will be enrolled in the case group of the present IR-CAD case-control study. Patients were diagnosed as IR-CAD if they have 1) evidence of rapidly progressive (occurred within 6 months or occurred on immunosuppressive therapy within 12 months of the last coronary revascularization) myocardial ischemia (typical symptoms and non-invasive evidence) despite standard treatment for secondary prevention of AS-CAD; 2) angiographic evidence of new coronary lesions (de novo stenosis or restenosis) considered to be relevant to myocardial ischemia; 3) evidence of inflammation (positive inflammation markers or established diagnosis of inflammatory diseases or use of immunosuppressive therapy). The comprehensive treatment for IR-CAD included: 1) intensified secondary prevention of AS-CAD; 2) immunosuppressive therapy; 3) coronary revascularization; 4) supportive therapies.

Patients who fulfill the inclusion/exclusion criteria for AS-CAD defined by the protocol of the present case-control study will be enrolled in the control group of the present case-control study. Patients will be diagnoses as AS-CAD if they 1) are ≥ 45 but < 65 years of age; 2) are receiving standard treatment for secondary prevention of AS-CAD after the last PCI which was performed 12±6 months ago; 3) do not have evidence of rapidly progressive (occurred within 6 months or occurred on immunosuppressive therapy within 12 months of the last PCI) myocardial ischemia (typical symptoms and non-invasive evidence); 4) do not have angiographic evidence of new coronary lesions (de novo stenosis or restenosis) considered to be relevant to myocardial ischemia.

Patients in the IR-CAD cohort study underwent examinations after they met the inclusion/exclusion criteria for IR-CAD based on a protocol specifically designed for the clinical management of IR-CAD patients. The results of the above examinations will be used as the examination results of the case group of the present IR-CAD case-control study. While patients in the control group of the present case-control study will undergo similar examinations after enrollment according to the protocol of the present case-control study.

The information regarding the baseline characteristics and the examination results, including demographics, clinical features, lab results, imaging findings, and prior treatment, will be collected and compared between the case group and the control group.

The primary endpoint is the rate of elevated erythrocyte sedimentation rate (ESR).

Eligible patients will be enrolled in the case group and the control group with a 2:1 ratio. The primary endpoint of the present case-control study is elevated erythrocyte sedimentation rate (ESR), which is defined as ESR > 15 mm for male, or ESR > 20 mm for female. In case of normal ESR, prior use of immunosuppressive therapy or prior diagnosis of autoimmune diseases before enrollment is regarded as the equivalent to elevated ESR. Based on currently available data from the IR-CAD cohort study, the rate of elevated ESR in the case group (IR-CAD patients) is 88.9% (8/9). The investigators hypothesize that the rate of elevated ESR in the control group (AS-CAD patients) is 20%. In consequence, 20 patients in the case group and 10 patients in the control group would be required to test the difference of the rate of the primary endpoint between the two groups at a significance level of 0.05 (α = 0.05) with a power of 90% (β = 0.10) and a drop-out rate of 20%.

Continuous variables will be presented as mean ± standard deviation (SD) or median (interquartile range [IQR]) and compared with two-sample t-test or Wilcoxon rank sum test, as appropriate. Categorical data will be demonstrated as n (%) and compared using Chi-square test or Fisher's exact test, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

Case group (IR-CAD patients):

1. 18 years of age or older, male or female.
2. Negative results of urine or blood pregnancy test for females with childbearing potential (not post-menopausal or surgically sterile).
3. Prior history of coronary revascularization (PCI or coronary artery bypass graft [CABG]).
4. Receiving standard treatment for secondary prevention of AS-CAD after the last coronary revascularization.
5. Hospitalization due to rapidly-progressive myocardial ischemia:

   * Typical symptoms of angina (Canadian Cardiovascular Society [CCS] III-IV) and non-invasive evidence of myocardial ischemia; and
   * Occurred within 6 months or occurred on immunosuppressive therapy within 12 months of the last coronary revascularization.
6. Angiographic evidence of new coronary lesions (de novo stenosis or restenosis) considered to be relevant to myocardial ischemia.
7. Evidence of inflammation:

   * At least one of the indexes indicating active inflammation has ever been elevated (ESR, high-sensitivity C-reactive protein [hs-CRP], interleukin [IL]-6, tumor necrosis factor [TNF]-α, ferritin, et al); or
   * Established diagnosis of systemic autoimmune disease or systemic vasculitis; or
   * Receiving immunosuppressive therapy.

Control group (AS-CAD patients):

1. ≥ 45 and < 65 years of age (based on the age distribution of the patients currently enrolled in the IR-CAD cohort study), male or female.
2. Negative results of urine or blood pregnancy test for females with childbearing potential (not post-menopausal or surgically sterile).
3. Currently, 12±6 months after the last PCI.
4. Receiving standard treatment for secondary prevention of AS-CAD after the last PCI.
5. Coronary angiography and/or optical coherence tomography (OCT) performed during the present hospitalization.
6. No evidence of rapidly-progressive myocardial ischemia, which is defined as follows:

   * Typical symptoms of angina (Canadian Cardiovascular Society [CCS] III-IV) and non-invasive evidence of myocardial ischemia; and
   * Occurred within 6 months or occurred on immunosuppressive therapy within 12 months of the last PCI.
7. No angiographic evidence of new coronary lesions (de novo stenosis or restenosis) considered to be relevant to myocardial ischemia.

Exclusion Criteria:

Case group (IR-CAD patients):

1. Coronary restenosis due to mechanical factors (stent under-expansion, stent mal-apposition, stent rupture, et al).
2. Other moderate to severe heart diseases (congenital heart disease, valvular heart disease, myocarditis, cardiomyopathy, pericardial diseases, pulmonary hypertension, heart failure, arrhythmia, et al).
3. Active acute or chronic infection (human immunodeficiency virus [HIV], tuberculosis, et al).
4. Active malignancy (diagnosed within 12 months or with ongoing requirement for treatment).
5. Vital organ failure.
6. Life expectancy < 1 year.
7. Contraindications for or intolerance to treatment for secondary prevention of AS-CAD, contrast agents, glucocorticoids, immunosuppressive agents.
8. In pregnancy or breast-feeding, or with intention to be pregnant during the study period.
9. Risk of non-compliance (history of drug addiction or alcohol abuse, et al).
10. Previous enrollment in this study.
11. Participation in another study within 30 days.
12. Involvement in the planning and conduct of this study (applying to investigators, contract research organization staffs, study site staffs, et al).
13. Any condition, which in the opinion of the investigators, would make it unsuitable for the patient to participate in this study.

Control group (AS-CAD patients):

The same as those for the case group (IR-CAD patients).

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The first 20 patients who were enrolled in the IR-CAD cohort study, which included patients who met the inclusion/exclusion criteria for IR-CAD and received comprehensive treatment, will be enrolled in the case group of the present IR-CAD case-control study.
  Patients who fulfill the inclusion/exclusion criteria for AS-CAD defined by the protocol of the present case-control study will be enrolled in the control group of the present case-control study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Elevated erythrocyte sedimentation rate (ESR) | From the last coronary revascularization up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with elevated ESR (> 15 mm for male or > 20 mm for female). In case of normal ESR, prior use of immunosuppressive therapy or prior diagnosis of autoimmune diseases before enrollment is regarded as the equivalent to elevated ESR.

SECONDARY OUTCOMES:
Age | On the day of enrollment.
  Age in years.
Female sex | On the day of enrollment.
  Percentage of patients with female sex.
Yellow race | On the day of enrollment.
  Percentage of patients with yellow race.
Acute coronary syndrome (ACS) | On the day of enrollment.
  Percentage of patients admitted due to ACS for the index hospitalization.
Chronic coronary syndrome (CCS). | On the day of enrollment.
  Percentage of patients admitted due to CCS for the index hospitalization.
Hypertension | On the day of enrollment.
  Percentage of patients with prior history of hypertension.
Dyslipidemia | On the day of enrollment.
  Percentage of patients with prior history of dyslipidemia.
Diabetes | On the day of enrollment.
  Percentage of patients with prior history of diabetes.
Smoking | On the day of enrollment.
  Percentage of patients with prior history of smoking.
Old myocardial infarction (OMI) | On the day of enrollment.
  Percentage of patients with prior history of OMI.
Percutaneous coronary intervention (PCI) | On the day of enrollment.
  Percentage of patients with prior history of PCI.
Coronary artery bypass graft (CABG) | On the day of enrollment.
  Percentage of patients with prior history of CABG.
Number of prior coronary revascularization | On the day of enrollment.
  Number of prior coronary revascularization
Blood pressure | On the day of enrollment.
  Measurement of blood pressure.
Heart rate | On the day of enrollment.
  Measurement of heart rate.
Body weight | On the day of enrollment.
  Measurement of body weight.
Height | On the day of enrollment.
  Measurement of height.
Body mass index (BMI) | On the day of enrollment.
  BMI = Body weight [kg] / (Height [m])^2
Antithrombotic agents | On the day of enrollment.
  Percentage of patients on antithrombotic agents.
β-blockers | On the day of enrollment.
  Percentage of patients on β-blockers.
Blood pressure-lowering agents | On the day of enrollment.
  Percentage of patients on blood pressure-lowering agents.
Lipid-lowering agents | On the day of enrollment.
  Percentage of patients on lipid-lowering agents.
Hypoglycemic agents | On the day of enrollment.
  Percentage of patients on hypoglycemic agents.
Glucocorticoids | On the day of enrollment.
  Percentage of patients on glucocorticoids.
Immunosuppressive agents | On the day of enrollment.
  Percentage of patients on immunosuppressive agents.
Other immunosuppressive therapy | On the day of enrollment.
  Percentage of patients on other immunosuppressive therapy.
Major adverse cardiovascular events (MACE) | From the last coronary revascularization up to the day of enrollment.
  Percentage of patients with death, or Q wave myocardial infarction, or unplanned myocardial ischemia-driven coronary revascularization (PCI or CABG), or unplanned myocardial ischemia-driven hospitalization.
Target vessel related major adverse cardiovascular events (TV-MACE) | From the last coronary revascularization up to the day of enrollment.
  Percentage of patients with cardiovascular death, or target vessel related Q wave myocardial infarction, or target vessel related unplanned myocardial ischemia-driven coronary revascularization (PCI or CABG), or target vessel related unplanned myocardial ischemia-driven hospitalization.
Hemoglobin | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of hemoglobin.
Red blood cell | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of red blood cell count.
White blood cell | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of white blood cell count.
Platelet | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of platelet count
Alanine aminotransferase (ALT) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of ALT.
Aspartate aminotransferase (AST) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of AST.
Gamma-glutamyl transferase (GGT) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of GGT.
Alkaline phosphatase (ALP) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of ALP.
Lactate dehydrogenase (LDH) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of LDH.
Total bilirubin (T-Bil) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of T-Bil.
Direct bilirubin (D-Bil) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of D-Bil.
Albumin | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of Albumin
Creatinine | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of creatinine.
Blood urea nitrogen (BUN) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of BUN.
Triiodothyronine (T3) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of T3.
Thyroxine (T4) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of T4.
Free triiodothyronine (FT3) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of FT3.
Free thyroxine (FT4) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of FT4.
Thyroid-stimulating hormone (TSH) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of TSH.
Total cholesterol (TC) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of TC.
Low-density lipoprotein cholesterol (LDL-C) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of LDL-C.
High-density lipoprotein cholesterol (HDL-C) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of HDL-C.
Triglyceride (TG) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of TG.
Apolipoprotein A (ApoA) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of ApoA.
Apolipoprotein B (ApoB) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of ApoB.
Lipoprotein (a) (Lp[a]) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of Lp(a).
Fasting blood glucose (FBG) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of FBG.
Hemoglobin A1c (HbA1c). | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of HbA1c.
Cardiac troponin I (cTnI) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of cTnI.
Creatine kinase-myocardial band (CK-MB) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of CK-MB.
Creatine kinase (CK) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of CK.
B-type natriuretic peptide (BNP) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of BNP.
N-terminal pro-B-type natriuretic peptide (NT-proBNP). | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of NT-proBNP.
Lupus anticoagulant | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of lupus anticoagulant.
Antiphospholipid antibody | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of antiphospholipid antibody.
Anti-phosphatidylserine antibody | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of anti-phosphatidylserine antibody.
Anti-prothrombin antibody | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of anti-prothrombin antibody.
Protein S | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of Protein S.
Protein C | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of Protein C.
Activated protein C resistance (APC-R) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of APC-R.
Anti-thrombin III | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of anti-thrombin III.
Maximum platelet aggregation (MPA) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of MPA.
Anti-nuclear antibody (ANA) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of ANA.
Anti-neutrophil cytoplasmic antibody (ANCA) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of ANCA.
Anti-endothelial cell antibody (AECA) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of AECA.
Rheumatoid factor (RF) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of RF.
Anti-cyclic citrullinated peptide (Anti-CCP) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of Anti-CCP.
Immunoglobulin | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of immunoglobulin.
Complement | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of complement.
Erythrocyte sedimentation rate (ESR) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of ESR.
High-sensitivity C-reactive protein (hs-CRP) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of hs-CRP.
Interleukin (IL)-6 | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of IL-6.
Tumor necrosis factor (TNF)-α. | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of TNF-α.
Pathological Q waves | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with pathological Q wave.
Dynamic ST-T changes | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with dynamic ST-T changes.
Segmental wall motion abnormality | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with segmental wall motion abnormality.
Left atrial diameter (LAD) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Measurement of LAD.
Left ventricular end-systolic diameter (LVESD) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Measurement of LVESD.
Left ventricular end-diastolic diameter (LVEDD) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Measurement of LVEDD.
Left ventricular ejection fraction (LVEF) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Measurement of LVEF.
Birmingham Vasculitis Activity Score (BVAS) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Result of BVAS (version 3) assessment.
Walking distance in 6 minutes | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Result of 6-minute walk test (6MWT).
Number of squats in 1 minute | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Result of 1-minute squatting test (1MST).
Temporal artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in either temporal artery on vascular ultrasound.
Carotid artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in either carotid artery on vascular ultrasound.
Vertebral artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in either vertebral artery on vascular ultrasound.
Subclavian artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in either subclavian artery on vascular ultrasound.
Iliac artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in either Iliac artery on vascular ultrasound.
Upper extremity artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in either upper extremity artery on vascular ultrasound.
Lower extremity artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in either lower extremity artery on vascular ultrasound.
Abdominal aorta stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in abdominal aorta on vascular ultrasound.
Celiac trunk stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in celiac trunk on vascular ultrasound.
Superior mesenteric artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in superior mesenteric artery on vascular ultrasound.
Renal artery stenosis | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Percentage of patients with ≥ 50% diameter stenosis in either renal artery on vascular ultrasound.
SYNTAX score | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Result of SYNTAX score assessment based on coronary angiogram.
Number of vessel segments with coronary lesions. | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Number of vessel segments with ≥ 50% diameter stenosis on coronary angiogram.
Target lesion minimal lumen area (TL-MLA) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Measurement of the minimum lumen area of the target lesion on optical coherence tomography (OCT).
Target lesion percent area stenosis (TL-%AS) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Measurement of percent area stenosis (% AS) of target lesion = { [ ( proximal RLA + distal RLA ) - (MLA × 2) ] / ( proximal RLA + distal RLA ) } × 100% in the cross-section with the MLA of the target lesion on optical coherence tomography (OCT). RLA = reference lumen area; MLA = minimum lumen area; % AS = percent area stenosis.

OTHER OUTCOMES:
Maximum standardized uptake value (SUVmax) | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  The mean of SUVmax of each major coronary artery on fibroblast activation protein inhibitor (FAPI) positron emission tomography/computed tomography (PET/CT).
RNA sequencing | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of RNA sequencing.
Proteomics | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of proteomics.
Metabolomics | From the index hospital admission up to 2 weeks of enrollment, but before the initiation of comprehensive treatment for patients with IR-CAD.
  Test result of metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Liu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Neumann FJ, Sousa-Uva M. 'Ten commandments' for the 2018 ESC/EACTS Guidelines on Myocardial Revascularization. Eur Heart J. 2019 Jan 7;40(2):79-80. doi: 10.1093/eurheartj/ehy855. No abstract available. PMID 30615155
- [Background] Fernandez DM, Giannarelli C. Immune cell profiling in atherosclerosis: role in research and precision medicine. Nat Rev Cardiol. 2022 Jan;19(1):43-58. doi: 10.1038/s41569-021-00589-2. Epub 2021 Jul 15. PMID 34267377
- [Background] Deroissart J, Porsch F, Koller T, Binder CJ. Anti-inflammatory and Immunomodulatory Therapies in Atherosclerosis. Handb Exp Pharmacol. 2022;270:359-404. doi: 10.1007/164_2021_505. PMID 34251531
- [Background] Engelen SE, Robinson AJB, Zurke YX, Monaco C. Therapeutic strategies targeting inflammation and immunity in atherosclerosis: how to proceed? Nat Rev Cardiol. 2022 Aug;19(8):522-542. doi: 10.1038/s41569-021-00668-4. Epub 2022 Jan 31. PMID 35102320
- [Background] Tucker B, Vaidya K, Cochran BJ, Patel S. Inflammation during Percutaneous Coronary Intervention-Prognostic Value, Mechanisms and Therapeutic Targets. Cells. 2021 Jun 4;10(6):1391. doi: 10.3390/cells10061391. PMID 34199975
- [Background] Kalkman DN, Aquino M, Claessen BE, Baber U, Guedeney P, Sorrentino S, Vogel B, de Winter RJ, Sweeny J, Kovacic JC, Shah S, Vijay P, Barman N, Kini A, Sharma S, Dangas GD, Mehran R. Residual inflammatory risk and the impact on clinical outcomes in patients after percutaneous coronary interventions. Eur Heart J. 2018 Dec 7;39(46):4101-4108. doi: 10.1093/eurheartj/ehy633. PMID 30358832
- [Background] Guedeney P, Claessen BE, Kalkman DN, Aquino M, Sorrentino S, Giustino G, Farhan S, Vogel B, Sartori S, Montalescot G, Sweeny J, Kovacic JC, Krishnan P, Barman N, Dangas G, Kini A, Baber U, Sharma S, Mehran R. Residual Inflammatory Risk in Patients With Low LDL Cholesterol Levels Undergoing Percutaneous Coronary Intervention. J Am Coll Cardiol. 2019 May 21;73(19):2401-2409. doi: 10.1016/j.jacc.2019.01.077. PMID 31097159
- [Background] Takahashi N, Dohi T, Endo H, Funamizu T, Wada H, Doi S, Kato Y, Ogita M, Okai I, Iwata H, Okazaki S, Isoda K, Miyauchi K, Shimada K. Residual Inflammation Indicated by High-Sensitivity C-Reactive Protein Predicts Worse Long-Term Clinical Outcomes in Japanese Patients after Percutaneous Coronary Intervention. J Clin Med. 2020 Apr 6;9(4):1033. doi: 10.3390/jcm9041033. PMID 32268533
- [Background] Kikuchi S, Okada K, Hibi K, Maejima N, Yabu N, Uchida K, Tamura K, Kimura K. Coronary arteritis: a case series. Eur Heart J Case Rep. 2020 Feb 17;4(2):1-6. doi: 10.1093/ehjcr/ytaa011. eCollection 2020 Apr. PMID 32352046
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; ESC Scientific Document Group. Fourth universal definition of myocardial infarction (2018). Eur Heart J. 2019 Jan 14;40(3):237-269. doi: 10.1093/eurheartj/ehy462. No abstract available. PMID 30165617
- [Background] Braunwald E. Unstable angina. A classification. Circulation. 1989 Aug;80(2):410-4. doi: 10.1161/01.cir.80.2.410. No abstract available. PMID 2752565